CLINICAL TRIAL: NCT03182556
Title: Comparison of the Efficacy of Electromyographic Biofeedback, Aerobic Exercise (Biodanza) and Stretching in Patients With Fibromyalgia.
Brief Title: Efficacy of Electromyographic Biofeedback, Aerobic Exercise and Stretching in Fibromyalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María del Mar Lopez-Rodriguez, Assistant Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mlr295
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Fibromyalgia
Keywords: Dance Therapy; Exercise; Myofeedback; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Biofeedback, Psychology; Aquatic Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stretching (Placebo Comparator): Stretching sessions was held twice a week in the University of Almería facilities, lasting approximately one hour and they included different muscle areas exercises as well as stretching across the board.
  Interventions: Behavioral: Electromyography-Biofeedback (EMG-BFB) training; Behavioral: Aquatic exercise
- Aquatic Exercise (Experimental): Aquatic Exercise program (Biodanza exercises) was carried out in a swimming-pool with a water temperature of approximately 29 ° C, preceded by a shower at a temperature of about 33-35 °C. Each session lasts an hour and they will held twice a week (Monday and Wednesday) during a period of time of three months (12 weeks).
  Interventions: Behavioral: Electromyography-Biofeedback (EMG-BFB) training
- Electromyography-Biofeedback training (Experimental): The whole treatment will last about 12 sessions. Each one lasts about 30 and 40 minutes and will be performed continuously once a week. The frequency may be increased if the level of tonic muscle tension becomes too high.
  Interventions: Behavioral: Aquatic exercise

INTERVENTIONS:
Behavioral: Electromyography-Biofeedback (EMG-BFB) training — The Chattanooga Intelect Advanced model was used with the surface EMG for 2 independent channels. The patient can observe on the screen as columns of varying their height in the function of the degree of muscular tension. Each session was configured as follows. First, a 2 minute period for adaptation and then we continue with a 2 minute period to establish the baseline. After that, a 7 minute training trial session to reduce the muscle tension as well as a pause of about 2 minutes. Then, it continued with two more trials of 7 minutes interleaved with another 2 minute break. Thus, the whole training lasts 29 minutes approximately. The pauses between the individual trials were intended to recover the baseline level to carry out a new trial which will start from a higher level of EMG.
  Other Names: Myofeedback; Surface electromyography biofeedback
  Arms: Aquatic Exercise; Stretching
Behavioral: Aquatic exercise — Aquatic Exercise program (Biodanza exercises) was carried out in a swimming-pool with a water temperature of approximately 29 ° C, preceded by a shower at a temperature of about 33-35 °C. Each session lasts an hour and they will held twice a week (Monday and Wednesday) during a period of time of three months (12 weeks).
  Other Names: Aquatic Biodanza; Aquatic Biodance; Aquatic aerobic exercise
  Arms: Electromyography-Biofeedback training; Stretching

SUMMARY:
Some authors claim that patients with musculoskeletal pain tend to underestimate their levels of muscle tension. The results of studies find evidences of the deficits in the perception of muscular tension in patients with chronic pain, being this the pathogenic factor in some musculoskeletal alterations. These studies show that patients with chronic pain can not identify their muscle tension and suggest that this contributes to maintaining pain. Thus, positive results have been found with relaxation and electromyographic biofeedback in patients with chronic pain. If these symptoms are due to excessive stress, patients should be able to benefit from regulation of muscle activity through BFB-EMG, thus learning to regulate the physiological variable. The study will be carried out in the electrotherapy laboratory of the Health Sciences Building of the University of Almeria. Initially, the sample will be chosen and the informed consent of the subjects will be obtained. Before the start of treatment, a baseline assessment of the dependent variables will be performed. Subsequently subjects will undergo three sessions of manipulative therapy over 12 weeks (one session per week). After the therapeutic intervention, a new determination of the dependent variables will be performed.

DETAILED DESCRIPTION:
Fibromyalgia (FM) affects nearly 2.4% of the Spanish population, mostly women aged between 40 and 60. This disease, which is characterized by a disturbance in their pain regulation with an increased sensitivity to painful stimuli and a decrease of pain threshold, has a strong impact on the patients' health and their quality of life, restricting the realization of their daily activities. Moreover, it presents a high prevalence of comorbidities, which increases the needs of these patients in terms of effective therapeutic management leading to higher health requirements.

In addition to that, FM response to drug treatments is low and its symptoms become more frequent simultaneously with adverse effects, and according to that, an individualized analysis becomes necessary as well as a multidisciplinary approach, since there is no absolute treatment up to now.

This study aims to compare the improvements obtained in the quality of life, pain and other FM symptoms respectively, by means of applying physical therapies (such as aerobic biodance exercise in aquatic environment and stretching exercises) and psychological treatments, such as electromyographic biofeedback (BFB-EMGS) based training.

Objectives:

To comparatively analyze the level of improvement that can be reached by FM patients, by means of pool exercises based treatments, stretching exercises and BFB-EMGS therapies.

Methodology:

The sample of this study consisted of FM diagnosed individuals who verified the following inclusion criteria:

* Aged over 18 years and below 69 years.
* FM diagnosed according to the American College of Rheumatology (ACR) criteria.
* To continue with their unchanged drug treatment for the duration of the study.
* To attend at least 60% of sessions to be considered to have completed both aquatic aerobic exercise treatment and stretching therapy, or to complete at least 12 sessions in the BFB-EMGS training case.

In addition to that, the exclusion criteria were:

* Aged over 69 years or below 18 years.
* To be involved in other non-pharmacological treatments.
* To display disorders such as heart, kidney or liver failures, which prevent the development of treatments.
* Other physical or mental disorders that could endanger the patient's health.
* Not have completed the minimum number of sessions of the corresponding therapy. Thus, this is an experimental study with randomized clinical trial design, consisting of three intervention groups, namely, aquatic aerobics group, stretching group and BFB-EMGS with stretching group. All groups were composed of 35 patients and were assessed before and after 12 weeks of treatment by a single investigator blinded to patient allocation.

Comparisons were established within each group, before and after 12 weeks of treatment (intragroup) and between groups (intergroup). In this way, all patient were asked to sign an informed consent and their demographics and health data were recorded in the first meeting.

Dependent variables.

* FM Impact Questionnaire (FIQ).
* McGill-Melzack questionnaire.
* Visual Analog pain Scale (VAS).
* The depression scale was estimated by means of the Center for Epidemiologic Studies Depression (CES-D).
* Pressure algometry.
* The anxiety was measured by the State Anxiety Inventory (SAI).
* The sleep quality was measured by the Pittsburgh Sleep Quality Index (PSQI).
* The number of tender points in each patient. Independent variables.
* Aerobic biodance program in pool;
* Stretching exercises program;
* BFB-EMGS training;

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 72 years and diagnosed with FMS according to 2010 ACR criteria. Before being included in the study, all the subjects must have signed an informed consent to ensure their participation, stating that it may be left at any time if were necessary.

Exclusion Criteria:

* Patients with physical or mental illness, infections, fever, hypotension, respiratory disorders which prevent the treatment realization, patients who do not maintain usual treatment during the study period or who do not perform the full intervention.

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-05-11 (Actual); Primary Completion 2013-04-17 (Actual); Study Completion 2016-09-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline Fibromyalgia Impact Questionnaire (FIQ) at 3 months. | At baseline and 12 weeks
  This questionnaire was designed to evaluate the influence of FMS in the patients' daily life. A properly validated Spanish version of FIQ was applied in this study.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI). | At baseline and 12 weeks
  This questionnaire consists of 19 items which allow evaluating the quality of sleep of the last month and differentiates between ''poor'' and ''good'' quality sleepers. The index is composed by seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction.
Center for Epidemiological Studies Depression Scale. | At baseline and 12 weeks
  A screening measure developed to identify current depressive symptomatology related to major or clinical depression in adults and adolescents.This questionnaire is a self-report inventory contains 20 items that are scored by respondents to indicate the frequency of symptoms during the previous week.
State-Trait Anxiety Inventory (STAI). | At baseline and 12 weeks
  This consists of 40 items which evaluate the state and the trait anxiety of a person.
Pressure algometry. | At baseline and 12 weeks
  The pressure algometer (Wagner FPI 10) is an instrument valid for the measurement and location of the pressure-sensitive points.
McGill Questionnaire. | At baseline and 12 weeks
  This questionnaire was designed and proposed by Melzack and Torgerson in order to quantify pain. Thus, it evaluates both quantitative and qualitative pain aspects.
Visual Analogical Scale (VAS). | At baseline and 12 weeks
  This scale was used to assess changes in pain intensity before and after treatment, and after each training session.

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Lopez-Rodriguez, PhD, Principal Investigator — Universidad de Almeria

IPD SHARING:
Plan to Share IPD: No